CLINICAL TRIAL: NCT03755687
Title: Effectiveness of Art Therapy Interventions for Adolescent Pain Management in the Pediatric Emergency Department
Brief Title: Art Therapy Pain Management Adolescents Pediatric ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: American Art Therapy Association (Unknown)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Associate Professor of Pediatrics in Emergency Medicine at CUMC, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS3531
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Pain
Keywords: Art Therapy; Pain Management; Pediatrics; Emergency Medicine
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Prospective observational pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Art Therapy Intervention (Experimental): Standardized mixed media art therapy directives (e.g. drawing/painting/collaging within a circle)
  Interventions: Other: Art Therapy Intervention

INTERVENTIONS:
Other: Art Therapy Intervention — Standardized mixed media art directives.

SUMMARY:
This project is studying adolescents between the ages of 12 to 18 years that come to the emergency department and are in pain. We want to find out how well art therapy is able to decrease the pain they are experiencing. Art therapy will involve making art and working with an art therapist to find new ways of expressing thoughts and feelings through art making.

In adolescents presenting to the emergency department with a painful condition, our aims are as follows:

Aim #1: To determine the degree that art therapy intervention reduces pain and anxiety.

Aim #2: To determine the degree that art therapy reduces pain and anxiety 1 hour after the intervention.

Aim #3: To explore the qualitative experience of patients undergoing art therapy intervention.

DETAILED DESCRIPTION:
Pain is one of the most common reasons for patients to visit the emergency department (ED), and can be treated using both complementary and pharmacological strategies. However, children are often undertreated for pain which results in not only short term problems, but long term consequences such as trauma and stress-induced disorders; health care avoidance as adults; increased pain sensitivity; and decreased response to future analgesia. There have been variable efforts made to improve the ED management of pain in children, but adolescents are frequently overlooked. A review of the literature revealed that art therapy for pain management in adolescents is understudied. The majority of studies describe the effects of art therapy on the emotional well-being in surgical and oncology populations in adults and children. The studies that did evaluate the effectiveness of art therapy for pain management in children focused primarily on surgical and medical oncology populations with children aged 2-14 years. Of these studies, none evaluated adolescents in the ED, which is a high volume and high stress environment that confers a distinct experience for patients compared to other medical settings. Evaluation of art therapy interventions using quantitative self-report measures with strong validity in children and further delineation of the patient experience related to art therapy is necessary. Advanced evaluation of aforementioned interventions would expand the evidence base needed to describe effectiveness of these interventions and support greater implementation and dissemination. These are the gaps in knowledge that the investigators aim to fill with the proposed study.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 18 years of age, inclusive
* Painful condition with self-reported pain score of >3/10

Exclusion Criteria:

* Critical illness as per attending physician
* Any neurological or developmental condition that precludes engagement in art therapy or ability to use a self-reported measure of pain
* Chronic disease associated with pain (e.g. sickle cell disease, fibromyalgia)
* Medical condition necessitating multiple painful procedures (e.g. malignancy, organ transplant)
* Does not speak English

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Change in patient pain intensity: Verbal Numerical Rating Scale | 1 hour
  Pain intensity measured using the Verbal Numerical Rating Scale. Minimum score (no pain) = 0, maximum score (most/worst pain) = 10.
Change in patient anxiety: Short Form STAI | 1 hour
  Anxiety measured using the short form State-Trait Anxiety Inventory (STAI). Consists of six short statements (e.g. "I feel calm", "I am tense"). For each statement, subject selects a response on a 4-point Likert scale, ranging from 1=Not at all, to 4=Very much.

SECONDARY OUTCOMES:
Perception of pain and anxiety: Qualitative questions | 1 hour
  Qualitative questions (3): 1. How would you describe this art therapy session? 2. What were some sensations you experienced in your body while you were engaged in the session? 3. Is there anything else you would like to say about what you are experiencing in your body and the art therapy session?

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Tsze, MD, MPH, Principal Investigator — Columbia University; Susanne M Bifano, MPS, MSED, Study Director — NewYork-Presbyterian Morgan Stanley Children's Hospital
Locations (1):
- NewYork Presbyterian Morgan Stanley Children's Hospital Emergency Department, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159